CLINICAL TRIAL: NCT04626128
Title: OASIS: Open-label, Dose-escalation, Phase 1/2a Study of the Safety and Tolerability of Suprachoroidally Administered CLS-AX Following Intravitreal Anti-VEGF Therapy in Subjects With Neovascular Age-related Macular Degeneration
Brief Title: Safety and Tolerability Study of Suprachoroidal Injection of CLS-AX Following Anti-VEGF Therapy in Neovascular AMD
Acronym: OASIS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clearside Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLS1002-101
Record Dates: First submitted 2020-11-02; First posted 2020-11-12 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: AMD; Wet-AMD; suprachoroidal; tyrosine kinase inhibitor; Microinjector; SCS
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: Four groups of approximately 5 participants are assigned to receive interventions in sequential dose escalation fashion based on prior milestones being reached.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Low Dose) (Experimental): Subjects will receive a low dose of 0.03 mg CLS-AX
  Interventions: Drug: CLS-AX; Drug: Anti-VEGF
- Cohort 2 (Low-mid Dose) (Experimental): Subjects will receive a low-mid dose of 0.10 mg CLS-AX
  Interventions: Drug: CLS-AX; Drug: Anti-VEGF
- Cohort 3 (High-mid Dose) (Experimental): Subjects will receive a high-mid dose of 0.50 mg CLS-AX
  Interventions: Drug: CLS-AX; Drug: Anti-VEGF
- Cohort 4 (High Dose) (Experimental): Subjects will receive a high-mid dose of 1.0 mg CLS-AX
  Interventions: Drug: CLS-AX; Drug: Anti-VEGF

INTERVENTIONS:
Drug: CLS-AX — injectable suspension of small molecule tyrosine kinase inhibitor (TKI)
  Other Names: axitinib injectable suspension
Drug: Anti-VEGF — Standard of care therapy used to block vascular endothelial growth factor
  Other Names: aflibercept (2mg)

SUMMARY:
To evaluate the safety and tolerability of suprachoroidally administered CLS-AX following intravitreal anti-VEGF therapy in subjects with neovascular age-related macular degeneration (AMD)

DETAILED DESCRIPTION:
Multi-center, open-label, dose-escalation, phase 1/2a, safety and tolerability study to evaluate four dose groups of suprachoroidally administered CLS-AX following intravitreal anti-VEGF therapy in up to a maximum of 25 subjects with neovascular age-related macular degeneration

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neovascular age-related macular degeneration in the study eye.
* Active subfoveal choroidal neovascularization (CNV) secondary to AMD
* Two or more prior anti-VEGF intravitreal injections
* EDTRS BCVA score ≤ 75 and ≥ 20 letters

Exclusion Criteria:

* Any active ocular disease, ocular disorders or conditions, prior ocular surgery or infection in the study eye other than nAMD
* Other than IVT anti-VEGF treatments, no topical ocular or intraocular or periocular corticosteroid, or other treatments for CNV
* IOP ≥ 25mmHg or cup-to-disc ratio >0.8
* Uncontrolled systemic disease (high risk or evidence of arterial and venous thromboembolism, CVA or stroke, unstable cardiovascular disease, uncontrolled hyperthyroidism, poor glycemic control, gastrointestinal bleed and/or high risk of GI perforation or fistula formation) or any other condition or therapy that would make the participant unsuitable for the study
* Currently enrolled in an investigational drug or device study or has used an investigational drug or device within 30 days or the Screening visit

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Coultas, PhD, Study Director — Clearside Biomedical, Inc.
Locations (11):
- United States (11):
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - California Retina Consultants, Bakersfield, California
  - Northern California Retina Vitreous Associates Medical Group, LLC, Mountain View, California
  - Retinal Consultants Medical Group, Sacramento, California
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Austin Retina Associates, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Consultants of Texas, San Antonio, Texas
  - Retina Consultants of Texas, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (Low-mid Dose) | Cohort 3 (High-mid Dose) | Cohort 4 (High Dose)
Started | 6 | 5 | 8 | 8
Safety Population (Defined as all enrolled participants who were administered CLS-AX, and from whom at least one post-Baseline safety measurement was obtained.) | 6 | 5 | 8 | 8
Pharmacokinetic Population (Defined as all participants that provide plasma samples for axitinib concentration analysis.) | 6 | 5 | 8 | 8
Completed | 6 | 4 | 8 | 8
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (Low-mid Dose) | Cohort 3 (High-mid Dose) | Cohort 4 (High Dose) | Total
Number analyzed (Participants) | 6 | 5 | 8 | 8 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.8 (11.55) | 78.2 (10.92) | 86.3 (6.48) | 76.5 (5.78) | 80.9 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5 | 5 | 15
  Male | 4 | 2 | 3 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 8 | 8 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 5 | 8 | 8 | 27
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 8 | 8 | 27
Duration of nAMD Diagnosis in the Study Eye [Mean (Standard Deviation); unit: months] | 50.13 (34.131) | 49.78 (21.905) | 66.64 (41.081) | 48.21 (48.045) | 54.39 (37.945)
Total Number of Prior nAMD Treatments in the Study Eye [Count of Participants; unit: Participants]
  0-2 injections | 0 | 0 | 0 | 0 | 0
  3-6 injections | 1 | 0 | 2 | 2 | 5
  7-12 injections | 0 | 1 | 0 | 1 | 2
  13-18 injections | 1 | 2 | 1 | 0 | 4
  >18 injections | 4 | 2 | 5 | 5 | 16
Pre injection Intraocular Pressure in the Study Eye at Baseline [Mean (Standard Deviation); unit: mmHg] — Intraocular pressure (IOP) is a diagnostic measurement of the fluid pressure, measured in millimeters of mercury, inside the eye. IOP was measured using Goldmann applanation tonometry or by use of a Tonopen tonometer. Normal eye pressure is usually considered to be between 10 and 20 mmHg (AAO.org). Untreated elevated eye pressure is a risk factor for glaucoma.
  mmHg | 15.3 (3.08) | 15.2 (2.39) | 13.3 (2.76) | 15.4 (3.81) | 14.7 (3.10)
Best Corrected Visual Acuity in the Study Eye at Baseline [Mean (Standard Deviation); unit: letters] — Best corrected visual acuity (BCVA) at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score attainable), with a higher score indicating better visual acuity.
  letters | 59.0 (16.43) | 65.6 (8.73) | 58.5 (13.69) | 65.8 (8.31) | 62.1 (12.06)
Central Subfield Thickness in the Study Eye at Baseline [Mean (Standard Deviation); unit: microns] — Central subfield thickness (CST) is a diagnostic measurement used in identifying the presence of edema in the circular area 1 mm in diameter centered around the fovea. CST was measured using spectral domain optical coherence tomography (SD-OCT). A central reading center graded the SD-OCT digital images. A negative change from baseline value represents a reduction in macular edema. Only images that were gradable by the central reading center were included in the analysis.
  microns | 231.2 (32.10) | 209.4 (17.39) | 202.0 (22.57) | 218.8 (40.01) | 214.8 (30.59)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with treatment-emergent adverse events (TEAEs) reported between the administration of CLS-AX and study exit.
Time Frame: Day 1 to Week 12
Population: Defined as all enrolled participants who were administered CLS-AX, and from whom at least one post-Baseline safety measurement was obtained.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (Low-mid Dose) | Cohort 3 (High-mid Dose) | Cohort 4 (High Dose)
Number analyzed (Participants) | 6 | 5 | 8 | 8
Participants | 1 | 2 | 1 | 3

2. Primary Outcome: Number of Participants With Serious Adverse Events
Description: Number of participants with serious adverse events (SAEs) reported between the administration of CLS-AX and study exit.
Time Frame: Day 1 to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (Low-mid Dose) | Cohort 3 (High-mid Dose) | Cohort 4 (High Dose)
Number analyzed (Participants) | 6 | 5 | 8 | 8
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Mean Change From Baseline in Pre Injection Intraocular Pressure (IOP)
Description: Intraocular pressure (IOP) is a diagnostic measurement of the fluid pressure, measured in millimeters of mercury, inside the eye. IOP was measured using Goldmann applanation tonometry or by use of a Tonopen tonometer. Normal eye pressure is usually considered to be between 10 and 20 mmHg (AAO.org). Untreated elevated eye pressure is a risk factor for glaucoma.
Time Frame: Weeks 4, 8 and 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (Low-mid Dose) | Cohort 3 (High-mid Dose) | Cohort 4 (High Dose)
Number analyzed (Participants) | 6 | 5 | 8 | 8
mmHg
  Week 4: number analyzed (Participants) | 6 | 5 | 7 | 8
  Week 4 | -2.8 (4.67) | -1.8 (4.15) | -0.3 (0.95) | 0.0 (4.66)
  Week 8: number analyzed (Participants) | 6 | 5 | 7 | 7
  Week 8 | -3.0 (3.16) | 0.6 (2.79) | 0.6 (1.90) | 1.6 (4.43)
  Week 12: number analyzed (Participants) | 6 | 4 | 8 | 8
  Week 12 | -3.0 (4.34) | 0.5 (1.91) | 0.9 (3.27) | 0.0 (3.38)

4. Secondary Outcome: Number of Participants Receiving Additional Intravitreal (IVT) Aflibercept Injections
Description: Number of participants receiving additional intravitreal aflibercept injections during the course of the study for nAMD. Participants qualified to receive additional IVT aflibercept injections based on protocol-defined criteria, including 1) loss of 10 or more letters in BCVA compared to the best prior study-assessed BCVA in the study eye that was attributed to intra- or sub-retinal fluid, 2) increase in central subfield thickness >75 microns from Baseline in the study eye, or 3) presence of vision-threatening hemorrhage due to AMD in the study eye. Additionally, a participant could receive additional IVT aflibercept injections in the study eye for reasons beyond the protocol-defined criteria if it was in the participant's best interest per the Investigator's judgment following best medical practice.
Time Frame: From Day 1 to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (Low-mid Dose) | Cohort 3 (High-mid Dose) | Cohort 4 (High Dose)
Number analyzed (Participants) | 6 | 5 | 8 | 8
Participants
  Week 4: number analyzed (Participants) | 6 | 5 | 7 | 8
  Week 4 | 0 | 1 | 1 | 4
  Week 8: number analyzed (Participants) | 6 | 5 | 7 | 7
  Week 8 | 4 | 2 | 1 | 1
  Week 12: number analyzed (Participants) | 6 | 4 | 8 | 8
  Week 12 | 1 | 2 | 1 | 1
  Day 1 to Week 12 | 4 | 4 | 2 | 4

5. Secondary Outcome: Number of Participants Qualifying to Receive Additional Intravitreal (IVT) Aflibercept Injections
Description: Number of participants qualifying to receive additional intravitreal aflibercept injections during the course of the study. Criteria included 1) loss of 10 or more letters in BCVA compared to the best prior study-assessed BCVA in the study eye that was attributed to intra- or sub-retinal fluid, 2) increase in central subfield thickness >75 microns from Baseline in the study eye, or 3) presence of vision-threatening hemorrhage due to AMD in the study eye.
Time Frame: Day 1 to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (Low-mid Dose) | Cohort 3 (High-mid Dose) | Cohort 4 (High Dose)
Number analyzed (Participants) | 6 | 5 | 8 | 8
Participants
  Week 4: number analyzed (Participants) | 6 | 5 | 7 | 8
  Week 4 | 0 | 1 | 1 | 3
  Week 8: number analyzed (Participants) | 6 | 5 | 7 | 7
  Week 8 | 4 | 2 | 1 | 0
  Week 12: number analyzed (Participants) | 6 | 4 | 8 | 8
  Week 12 | 1 | 2 | 2 | 2
  Day 1 to Week 12 | 4 | 4 | 2 | 3

6. Secondary Outcome: Mean Change From Baseline (Visit 2) in Central Subfield Thickness (CST) in the Study Eye
Description: Central subfield thickness (CST) is a diagnostic measurement used in identifying the presence of edema in the circular area 1 mm in diameter centered around the fovea. CST was measured using spectral domain optical coherence tomography (SD-OCT). A central reading center graded the SD-OCT digital images. A negative change from baseline value represents a reduction in macular edema. Only images that were gradable by the central reading center were included in the analysis.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (Low-mid Dose) | Cohort 3 (High-mid Dose) | Cohort 4 (High Dose)
Number analyzed (Participants) | 6 | 5 | 8 | 8
microns
  Week 4: number analyzed (Participants) | 6 | 5 | 7 | 8
  Week 4 | 22.3 (23.46) | 22.0 (17.83) | 21.1 (22.62) | 26.6 (26.45)
  Week 8: number analyzed (Participants) | 6 | 5 | 7 | 7
  Week 8 | 62.8 (57.60) | 21.8 (32.58) | 21.9 (25.75) | 9.9 (17.87)
  Week 12: number analyzed (Participants) | 6 | 4 | 8 | 8
  Week 12 | 8.8 (14.50) | 45.8 (69.72) | 29.1 (37.89) | 18.6 (27.33)

7. Secondary Outcome: Mean Change From Baseline (Visit 2) in Best Corrected Visual Acuity (BCVA) Letter Score in the Study Eye
Description: BCVA measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting test distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score attainable), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (Low-mid Dose) | Cohort 3 (High-mid Dose) | Cohort 4 (High Dose)
Number analyzed (Participants) | 6 | 5 | 8 | 8
letters
  Week 4: number analyzed (Participants) | 6 | 5 | 7 | 8
  Week 4 | 4.7 (3.78) | 0.2 (1.64) | -0.6 (4.61) | 1.0 (2.20)
  Week 8: number analyzed (Participants) | 6 | 5 | 7 | 7
  Week 8 | -0.2 (7.41) | -3.6 (2.30) | 0.6 (5.83) | 1.6 (2.94)
  Week 12: number analyzed (Participants) | 6 | 4 | 8 | 8
  Week 12 | 2.2 (4.92) | -6.3 (9.18) | -2.1 (4.45) | 0.3 (3.28)

8. Secondary Outcome: Maximum Plasma Concentration [Cmax] of Axitinib
Description: Maximum (or peak) plasma concentration of axitinib during the course of the study. Plasma samples were collected pre-dose at Baseline, 60 minutes post-dose at Baseline, and at Weeks 4 and 12. Peak quantifiable levels, based on a lower level of quantitation (LLOQ) of 0.01 ng/mL, were included in the analysis.
Time Frame: Day 1 to Week 12
Population: Defined as all participants that provide plasma samples for axitinib concentration analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (Low-mid Dose) | Cohort 3 (High-mid Dose) | Cohort 4 (High Dose)
Number analyzed (Participants) | 6 | 5 | 8 | 8
ng/mL | 0.0101 (0.00949) | 0.0264 (0.0242) | 0.0749 (0.111) | 0.0602 (0.0251)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 12 weeks following CLS-AX administration.
Arm/Group | Cohort 1 (Low Dose) | Cohort 2 (Low-mid Dose) | Cohort 3 (High-mid Dose) | Cohort 4 (High Dose)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/6 | 2/5 | 1/8 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Low Dose) (N=6) | Cohort 2 (Low-mid Dose) (N=5) | Cohort 3 (High-mid Dose) (N=8) | Cohort 4 (High Dose) (N=8)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Study eye
Conjunctival oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Study eye
Macular degeneration (Eye disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) — Study eye
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information concerning CLS1002-101 and the operations of Clearside Biomedical, Inc. are considered CONFIDENTIAL and shall remain the sole property of Clearside Biomedical Inc. The institutions and Investigators participating in this study shall have no right to publish or present the results of this study without the prior written consent of Clearside Biomedical, Inc.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT04626128/Prot_SAP_000.pdf